CLINICAL TRIAL: NCT03518411
Title: Adaptation of the One-session CBT Protocol for Prevention of Mental Illness for Brazilian Portuguese: Open Clinical Trial
Brief Title: Adaptation of the One-session CBT Protocol for Prevention of Mental Illness for Brazilian Portuguese
Acronym: UP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mariane Bagatin Bermudez (Other)
Responsible Party: Sponsor-Investigator, Mariane Bagatin Bermudez, MD, Hospital de Clinicas de Porto Alegre
Organization: Hospital de Clinicas de Porto Alegre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 73658817.3.1001.5327
Record Dates: First submitted 2017-12-14; First posted 2018-05-08 (Actual); Last update posted 2018-05-08 (Actual); Status verified 2018-05

CONDITIONS: Mental Disorder; CBT
MeSH Terms: conditions — Mental Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Medical Students (Experimental): Cognitive Behavioral Therapy Protocol
  Interventions: Other: Cognitive Behavioral Therapy

INTERVENTIONS:
Other: Cognitive Behavioral Therapy — One-Session Unified Protocol

SUMMARY:
1. Recruitment of medicine students of federal university.
2. Psychiatric interview (MINI) and sclaes application.
3. Protocol of CBT
4. Scales and MINI will be applied at the times of 7, 30 and 90 days after the end of the therapy.
5. Statistical analysis

ELIGIBILITY:
Inclusion Criteria:

* be medical student
* be over 18 years of age
* agree to the Term of Free and Informed Consent.

Exclusion Criteria:

* Students with psychotic illness, severe depression, manic episode or acute psychiatric risk.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-11-30 (Estimated)

PRIMARY OUTCOMES:
Prevention of anxiety symptoms | 90 days after
  Overall Anxiety Severity and Impairment Scale (OASIS). It is a 5-item self-report measure that can be used to assess severity and impairment associated with any anxiety disorder. Respondents select among five different response options for each item, which are coded 0-4 and summed to obtain a total score. A cut-score of 8 correctly classified 87% of this sample as having an anxiety diagnosis or not.

SECONDARY OUTCOMES:
Prevention of depression symptoms | 90 days after
  Beck Depression Inventory (BDI). It is a 21-question multiple-choice self-report inventory for measuring the severity of depression. Each question had a set of at least four possible (0 to 3) responses, ranging in intensity. Scores: 0-9: indicates minimal depression, 10-18: indicates mild depression, 19-29: indicates moderate depression, 30-63: indicates severe depression.

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Blaya, Study Director — Hospital de Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fisak BJ Jr, Richard D, Mann A. The prevention of child and adolescent anxiety: a meta-analytic review. Prev Sci. 2011 Sep;12(3):255-68. doi: 10.1007/s11121-011-0210-0. PMID 21437675
- [Background] Goebert D, Thompson D, Takeshita J, Beach C, Bryson P, Ephgrave K, Kent A, Kunkel M, Schechter J, Tate J. Depressive symptoms in medical students and residents: a multischool study. Acad Med. 2009 Feb;84(2):236-41. doi: 10.1097/ACM.0b013e31819391bb. PMID 19174678
- [Background] Guille C, Zhao Z, Krystal J, Nichols B, Brady K, Sen S. Web-Based Cognitive Behavioral Therapy Intervention for the Prevention of Suicidal Ideation in Medical Interns: A Randomized Clinical Trial. JAMA Psychiatry. 2015 Dec;72(12):1192-8. doi: 10.1001/jamapsychiatry.2015.1880. PMID 26535958
- [Background] Rotenstein LS, Ramos MA, Torre M, Segal JB, Peluso MJ, Guille C, Sen S, Mata DA. Prevalence of Depression, Depressive Symptoms, and Suicidal Ideation Among Medical Students: A Systematic Review and Meta-Analysis. JAMA. 2016 Dec 6;316(21):2214-2236. doi: 10.1001/jama.2016.17324. PMID 27923088
- [Result] Bentley KH, Boettcher H, Bullis JR, Carl JR, Conklin LR, Sauer-Zavala S, Pierre-Louis C, Farchione TJ, Barlow DH. Development of a Single-Session, Transdiagnostic Preventive Intervention for Young Adults at Risk for Emotional Disorders. Behav Modif. 2018 Sep;42(5):781-805. doi: 10.1177/0145445517734354. Epub 2017 Oct 13. PMID 29029563